CLINICAL TRIAL: NCT06714409
Title: A Parallel-group, Single-center, Two-arm Treatment Study to Assess the Safety and Effectiveness of Venous Ultrasound Guided Decongestion in Adult Patients Hospitalized with Acute Decompensated Heart Failure.
Brief Title: Venous Ultrasound Guided Organ Decongestion in Patients Hospitalized with Acute Decompensated Heart Failure
Acronym: VExOUS-ADHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Bård Waldum-Grevbo, Medical professor, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 744207
Record Dates: First submitted 2024-11-21; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Cardiorenal Syndrome; Heart Failure; Acute Kidney Injury; Acute Decompensated Heart Failure
Keywords: Cardiorenal syndrome; Acute kidney injury; Heart failure; VExUS; Venous congestion
MeSH Terms: conditions — Cardio-Renal Syndrome; Heart Failure; Acute Kidney Injury; Hyperemia

STUDY DESIGN:
Intervention Model Description: Single centre, parallel group, randomized controlled trail. Approximately 250 participants will be screened to achieve 90 randomly enrolled to study intervention and 90 participants to SOC arm for an estimated total of 180 evaluable participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Patients in the intervention arm will undergo VExUS examinations at 1st day of inclusion, every other day while hospitalized and at discharge. The results from the VExUS examination (VExUS score) will be provided to the treatment team and the treatment team decides the individual treatment regime based on available information, with the overall goal to optimize decongestionand HF treatment according to current hospital standards. Safety issues and AEs will be assessed.In both gropus echocardiography will be performed at least once during the hospital stay.
  Interventions: Diagnostic Test: VExUS guided decongestion
- Standard of care (No Intervention): Patients will undergo VExUS examinations at 1st day of inclusion and at discharge. The results from the VExUS examinations (VExUS score) will NOT be provided to the treatment team. They will be treated and followed up according to standard of care. In both gropus echocardiography will be performed at least once during the hospital stay.

INTERVENTIONS:
Diagnostic Test: VExUS guided decongestion — Treatment team will be provided information about venous organ congestion status.
  Arms: Intervention arm

SUMMARY:
The purpose of this study is to assess the feasibility, safety and effectiveness of VExUS guided organ decongestion compared to standard of care in patients hospitalized with acute decompensated heart failue (ADHF).

180 patients will be randomly assigned to either intervention (VExUS) arm or standard of care (SOC) arm. In the intervention arm, the treatment team will be informed by the study team about the results of the VExUS examination to supplement the clinical decision of proper decongestion treatment, while no information will be provided in the standard of care arm. Study visits are scheduled every second day while hospitalized, end of study is set to day of discharge from the ward. Telephone consultation and review of medical journal scheduled after 6 months to assess exploratory endpoints.

The overall rationale of the the study is to investigate if venous organ congestion investigated by VExUS score, is a modifiable risk factor in patients hospitalized with ADHF. And secondary to assess if venous organ decongestion guided by VExUS score may safely be implemented in patients hospitalized with ADHF and result in:

* differences in length of hospitalization
* changes in biomarkers of cardiac strain
* changes in renal function and markers of renal injury
* achieved doses of heart failure treatment at discharge
* in-hospital complications

Safety measures with special attention on symptomatic hypotension, arrhythmias, metabolic alkalosis and electrolyte disturbances will be addressed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above
* Admitted the ward of Department of Cardiology OUH Ullevål with a clinical diagnosis of ADHFdefined by European Society of Cardiology
* Pro-BNP > 800 ng/l at first day of admission
* Capable of giving signed informed consent

Exclusion Criteria:

- Any medical or psychiatric condition which in the opinion of the investigatorprecludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in VExUS score | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  The findings from Doppler ultrasonography of the hepatic vein, portal vein, and interlobar renal vein will be graded using the VExUS score, which reflects the degree of venous congestion. The scale ranges from 0 to 3, where a score of 0 indicates no signs of congestion, 1 indicates mild congestion, 2 indicates moderate congestion, and 3 indicates severe congestion.

SECONDARY OUTCOMES:
Change in NT-ProBNP | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Change in biomarker NT-ProBNP in serum.
Change in estimated renal glomerular filtration rate | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Estimated glomerular filtration rate (eGFR) is calculated based on serum creatinine, age and gender.
Change in urine albumin creatinine ratio | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Urine albumin creatinine is measured in spot urine sample.
Change in symptoms | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Participants are asked to grade their symptoms using a 7-point Likert scale ranging from 1 to 7, where 1 indicates markedly better, 4 indicates no change, and 7 indicates markedly worse. Additionally, participants are asked to report their general condition and level of dyspnea on a Visual Analogue Scale (VAS) where 0 is negative and 100 is positive.
Length of hospitalization | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Number of days from inclusion to discharge from hospital.
Achieved dosage of HF medications at discharge | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Current heart failure medication compared to target dose in the national recommendations of HF-patient population.
Safety | From the time of enrollment until hospital discharge, typically ranging from 3 to 21 days.
  Rates of symptomatic hypotension,worsening renal function, arrhythmias, severe metabolic alkalosis and electrolyte disturbances

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Longino A, Martin K, Leyba K, Siegel G, Thai TN, Riscinti M, Douglas IS, Gill E, Burke J. Prospective Evaluation of Venous Excess Ultrasound for Estimation of Venous Congestion. Chest. 2024 Mar;165(3):590-600. doi: 10.1016/j.chest.2023.09.029. Epub 2023 Oct 7. PMID 37813180
- [Background] Damman K, van Deursen VM, Navis G, Voors AA, van Veldhuisen DJ, Hillege HL. Increased central venous pressure is associated with impaired renal function and mortality in a broad spectrum of patients with cardiovascular disease. J Am Coll Cardiol. 2009 Feb 17;53(7):582-588. doi: 10.1016/j.jacc.2008.08.080. PMID 19215832
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Taylor DO, Starling RC, Young JB, Tang WHW. Importance of venous congestion for worsening of renal function in advanced decompensated heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):589-596. doi: 10.1016/j.jacc.2008.05.068. PMID 19215833
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297